CLINICAL TRIAL: NCT01100164
Title: A Phase III, Non-inferiority, Double-blind, Unicenter Clinical Trial With Two Treatment Arms - Test Group With Eszopiclone 3 mg Versus Zopiclone 7.5 mg - for the Treatment of Insomnia
Brief Title: A Non-inferiority Study With Two Treatment Arms Eszopiclone 3 mg Versus Zopiclone 7.5 mg - for the Treatment of Insomnia
Acronym: Eszo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EF097
Record Dates: First submitted 2010-04-05; First posted 2010-04-08 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2010-03

CONDITIONS: INSOMNIA
Keywords: INSOMNIA; FOR THE TREATMENT OF INSOMNIA
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone; zopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- eszopiclone 3 mg (Experimental): Eszopiclone - once a day (30 minutes before lying down to sleep for a period of 4 weeks of treatment)
  Interventions: Drug: Eszopiclone
- zopiclone 7,5mg (Active Comparator): Zopiclone once a day (30 minutes before lying down to sleep for a period of 4 weeks of treatment)
  Interventions: Drug: Zopiclone

INTERVENTIONS:
Drug: Eszopiclone — Eszopiclone - once a day (30 minutes before lying down to sleep for a period of 4 weeks of treatment)
  Arms: eszopiclone 3 mg
Drug: Zopiclone — Zopiclone - once a day (30 minutes before lying down to sleep for a period of 4 weeks of treatment)
  Arms: zopiclone 7,5mg

SUMMARY:
The primary objective of the study is to determine whether eszopiclone (Eurofarma) is non-inferior to the reference drug zopiclone (Imovane®, Sanofi-Aventis) in the treatment of insomnia.

DETAILED DESCRIPTION:
The primary objective of the study is to determine whether eszopiclone (Eurofarma) is non-inferior to the reference drug zopiclone (Imovane®, Sanofi-Aventis) in the treatment of insomnia. To that end, the latency to persistent sleep (LPS) will be used as a primary endpoint at the end of the treatment, measured by polysomnography.

The secondary objectives and endpoints of this study are as follows:

* To evaluate the efficiency of eszopiclone compared to zopiclone by means of the patient's clinical history, using as secondary endpoints:
* Variables of the sleep diary of the Associação Fundo de Incentivo à Psicofarmacologia (see Appendix A), namely:
* Latency time to the beginning of the sleep;
* Frequency of night wake-ups;
* Time awake during bedtime;
* Early morning awakening;
* Total time in bed;
* Sleep efficiency;
* Sleep variables measured by actigraph;
* Insomnia Severity Index (see Appendix B);45
* Pittsburgh Sleep Quality Index (see Appendix C);46
* To evaluate the safety of eszopiclone compared to zopiclone by means of adverse events in each study arm.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form for the study;
* Be ≥ 20 to ≥ 64 years old;
* Have diagnosis of symptomatic primary insomnia for at least 3 months;
* Have polysomnography conducted at least 90 days before the inclusion in the study with sleep time less than 6.5 hours and sleep latency ≥ 20 minutes;
* Be able not to take any insomnia medication for 14 days before randomization to the study (washout period).

Exclusion Criteria:

* Diagnosis of other sleep disorder by polysomnography conducted 90 days before the inclusion in the study;
* Use of any medication affecting the sleep, such as psychotropic, hypnotic or antihistamine agents for at least 15 days before the inclusion in the study;
* Use of any herbal supplement for insomnia or melatonin during the 14 days before entering the study;
* Current use of liver metabolized medication, especially those metabolized through the cytochrome P450 enzyme complex, especially through the CYP3A4 and/or CYP2E1 routes;
* History of daily use of alcohol beverages in quantities equivalent - from the ethanol standpoint - to two cans of beer a day (35 g of alcohol/day);
* History of substance abuse or dependence;
* Patients with severe co-morbidities (at the investigator's opinion);
* Presence of liver disorders, cirrhosis or liver failure;
* Presence of psychiatric disorders diagnosed at the adult life or currently under treatment;
* Pregnant and breastfeeding women and women who want to become pregnant during the study period and who refuse to use a proper contraceptive methods during the study.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 263 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Latency to persistent sleep measured by polysomnography | 4 weeks
  Determine whether eszopiclone is noninferior to the reference drug zopiclone (Imovane®) in the treatment of insomnia. The latency to persistent sleep will be used as a primary endpoint at the end of the treatment, measured by polysomnography

SECONDARY OUTCOMES:
Efficiency using the variables latency time to persistent sleep, frequency of night awakenings, time awake during bedtime, early morning awakening, total time in bed, total time awake and sleep efficiency | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CRDB - Clinical Research & Development Brazil, São Paulo, Brazil

REFERENCES:
- [Derived] Pinto LR Jr, Bittencourt LR, Treptow EC, Braga LR, Tufik S. Eszopiclone versus zopiclone in the treatment of insomnia. Clinics (Sao Paulo). 2016 Jan;71(1):5-9. doi: 10.6061/clinics/2016(01)02. PMID 26872077